CLINICAL TRIAL: NCT03429608
Title: Quantitative Estimation of Thrombus Burden in Patients With ST Elevation Acute Myocardial Infarction (STEMI) With the Use of Micro-computed Tomography-A Methodological Approach (QUEST-STEMI)
Brief Title: Quantitative Estimation of Thrombus Burden in Patients With STEMI Using Micro-Computed Tomography (QUEST-STEMI)
Acronym: QUEST-STEMI
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Hellenic Centre for Marine Research (Unknown); Harvard Medical School (HMS and HSDM) (Other); MHAT Hadji Dimitar Hospital, Sliven, Bulgaria (Unknown)
Responsible Party: Principal Investigator, Karagiannidis Efstratios, MD, MSc, Phd candidate, Aristotle University Of Thessaloniki
Other Study IDs: 20170210
Record Dates: First submitted 2018-01-25; First posted 2018-02-12 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: ST Elevation Myocardial Infarction; Thrombi
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — aspirated thrombi from patients with ST elevation myocardial infarction, who undergo primary PCI and thrombus aspiration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with low thrombus burden: patients with the lower volume of aspirated thrombi, as measured using micro-CT
- patients with high thrombus burden: patients with the higher volume of aspirated thrombi, as measured using micro-CT

SUMMARY:
The study aims to assess for the first time, through the application of innovative technologies (micro-CT), important characteristics of aspirated thrombi (such as their volume and their density), which might be linked to certain clinical outcomes, in patients presenting with STEMI and referred for primary Percutaneous Coronary Intervention (PCI). To this end, a methodology for the exact estimation of thrombus burden by measuring the volume and the density of aspirated thrombi will be developed. After being aspirated using dedicated catheters, thrombi will be preserved in formalin and their volume and their density will be calculated with the use of micro-CT. Having a better resolution than conventional computed tomography, micro-CT will allow us to create 3D models of aspirated thrombi from a series of x-ray projection images. These 3D models will be further analyzed in order to find the volume and the density of aspirated thrombi. Shape analysis of the surface of aspirated thrombi and potential differences in their structure will also be assessed. Correlation of these variables with clinical parameters and angiographic outcomes will be attempted.

Thus, a risk-stratification model will be developed combining:

* Clinical and laboratory data,
* Angiographic parameters,
* Data regarding the volume, the density and the composition of aspirated thrombi.

This model will enable the stratification of the cardiovascular and cerebrovascular risk of patients and the identification of who will benefit from thrombus aspiration, providing a personalized approach in treating patients with STEMI.

DETAILED DESCRIPTION:
Acute myocardial infarction with ST elevation (STEMI) remains one of the leading causes of mortality in developed countries, in spite of the important advances in pharmacological therapy and in mechanical reperfusion therapy. Having an important role in provoking ischemia, thrombus has been studied in many clinical trials and high thrombus burden has been proven to be an independent risk factor for stent thrombosis and for Major Adverse Clinical outcomes. However large randomized controlled trials concerning thrombus aspiration showed controversial results, providing as a whole no evidence of distinct benefits for thrombus aspiration. A possible explanation could be that aspiration was performed as a routine strategy in all of these trials, whereas these patients should be considered as a heterogeneous group and thus they should be risk-stratified. For this reason, it is of paramount importance to classify patients according to the volume of thrombus burden. The currently existing classifications of thrombus burden (the most important being those of Gibson and of Sianos) are based on visual assessment of angiographic characteristics and thus they are not reflecting the volume of the thrombi in actual, absolute numbers.

The main purpose of the study is to develop a methodology for the exact estimation of thrombus burden by measuring the volume and the density of aspirated thrombi in patients presenting with STEMI and referred for primary PCI. After being aspirated using dedicated catheters, thrombi will be preserved in formalin and their volume will be calculated with the use of micro-CT. The scanning procedure results into a series of projection images arranged in the form of image stacks which, in turn, are reformed in sections (cross section images) with the use of the NRecon (Bruker, Kontich, Belgium) software, which applies a modified algorithm of backward projection Feldkamp. The resulting sections will be combined to create the 3D models which will be further analyzed to extract useful measurements for the characteristics of the thrombi, such as for the volume and the elative density. Shape analysis on the surface and internal structure of the three-dimensional representations of the specimens will lead to the identification of the important features that can be used to estimate variability within samples and perform clustering for the significant differences between clots. In addition, possible differences in clot internal and external structure (e.g. architecture of the various cell types) will be assessed through the 3D models rendered from the stacks of images The Secondary end points of the study include the examination of the association of the aforementioned variables with the angiographic classification of thrombus burden (according to Sianos), with electrocardiographic and angiographic characteristics suggestive of poor patient prognosis and with major adverse cardiac events during the follow-up period of one year.

This method could become the gold standard for the exact measurement of thrombus burden and could be used in larger, clinically-oriented trials to help stratify patients with thrombus burden according to their risk for adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with symptoms of myocardial ischemia lasting for more than 30 minutes
* Definite ECG changes indicating STEMI
* Patients undergoing primary PCI within 12 hours from symptom onset
* Possibility to perform thrombus aspiration
* Age>18 years
* Written informed consent prior to enrolment in the clinical trial

Exclusion Criteria:

* Treatment with fibrinolytic therapy for qualifying index STEMI event
* Patients with known intolerance to aspirin, ticagrelor or heparin
* Patients with active internal bleeding
* Patients with a recent history of intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients presenting with ST elevation myocardial infarction, who undergo primary PCI and thrombus aspiration
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
volume of aspirated thrombus burden | 12 months
  The volume of aspirated thrombi will be quantified using micro-CT.
density of aspirated thrombus burden | 12 months
  The density of aspirated thrombi will be quantified using micro-CT.
MACCE-free survival | 12 months
  Time between the date of diagnosis and MACCE during the follow-up period of 12 months. MACCE are defined as any of the following: cardiac death, cerebrovascular death, acute myocardial infarction, target lesion revascularization, stent thrombosis or stroke.

SECONDARY OUTCOMES:
association between thrombus volume with factors from patients medical history | 12 months
  Potential association of thrombus volume (as assessed using micro-ct) with factors potentially affecting thrombus burden, including history of diabetes mellitus (dichotomous variable yes/no), use of antiplatelet drugs or anticoagulants (dichotomous variable yes/no),pain-to-balloon time (in minutes) and history of smoking (dichotomous variable yes/no) will be explored and reported.
association between thrombus density with factors from patients medical history | 12 months
  Potential association of thrombus density ( as assessed using micro-CT) with factors potentially affecting thrombus burden, including history of diabetes mellitus (dichotomous variable yes/no), use of antiplatelet drugs or anticoagulants (dichotomous variable yes/no),pain-to-balloon time (in minutes) and history of smoking (dichotomous variable yes/no) will be explored and reported.
Correlation of the volume of aspirated thrombus burden with the Sianos' classification of thrombus burden | 12 months
  Potential correlation of the volume of aspirated thrombus burden, as assessed using the micro-CT and the angiographic classification of thrombus burden according to Sianos will be explored. According to Sianos' classification thrombi are classified in the following categories: G0,G1,G2,G3,G4.
Correlation of thrombus density with the Sianos' classification of thrombus burden | 12 months
  Potential correlation of thrombus density, as assessed using the micro-CT and the angiographic classification of thrombus burden according to Sianos will be explored.
association of thrombus volume with electrocardiographic outcomes suggestive of poor patient prognosis | 12 months
  Potential association of thrombus volume as measured using micro-CT with ST segment resolution will be explored. ST resolution will be classified as complete (>70%), partial (30-70%), or absent (<30%).
association of thrombus density with electrocardiographic outcomes suggestive of poor patient prognosis | 12 months
  Potential association of thrombus density as measured using micro-CT with ST segment resolution will be explored. ST resolution will be classified as complete (>70%), partial (30-70%), or absent (<30%).
association of thrombus volume with post-procedural Thrombolysis in Myocardial Infarction(TIMI) flow | 12 months
  Potential association of thrombus volume as measured using micro-CT, with post-procedural TIMI flow (classified as previously described: TIMI flow 0,1,2 or 3) will be explored
association of thrombus density with post-procedural TIMI flow | 12 months
  Potential association of thrombus density as measured using micro-CT, with post-procedural TIMI flow (classified as previously described: TIMI flow 0,1,2 or 3) will be explored
association of thrombus volume with myocardial blush grade | 12 months
  Potential association of thrombus volume as measured using micro-CT, with myocardial blush grade (classified as previously described: myocardial blush grade 0, myocardial blush grade 1, myocardial blush grade 2 and myocardial blush grade 3) will be explored.
association of thrombus density with myocardial blush grade | 12 months
  Potential association of thrombus density as measured using micro-CT, with myocardial blush grade (classified as previously described: myocardial blush grade 0, myocardial blush grade 1, myocardial blush grade 2 and myocardial blush grade 3) will be explored.
association of thrombus volume with distal embolization . | 12 months
  Potential association of thrombus volume as measured using micro-CT, with distal embolization (dichotomous variable yes/no) will be explored.
association of thrombus density with distal embolization . | 12 months
  Potential association of thrombus density as measured using micro-CT, with distal embolization (dichotomous variable yes/no) will be explored.
association of thrombus volume with Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 12 months
  Potential association of thrombus volume, as measured using micro-CT with MACCE during the follow-up period of 12 months, will be explored. MACCE are defined as any of the following: cardiac death, cerebrovascular death, acute myocardial infarction, target lesion revascularization, stent thrombosis or stroke.
association of thrombus density with Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 12 months
  Potential association of thrombus density, as measured using micro-CT with MACCE during the follow-up period of 12 months, will be explored. MACCE are defined as any of the following: cardiac death, cerebrovascular death, acute myocardial infarction, target lesion revascularization, stent thrombosis or stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Sianos, MD,PhD, FESC, Study Chair — Associate Professor of Cardiology, School of Medicine, Aristotle University of Thessaloniki; Efstratios Karagiannidis, MD,MSc, Principal Investigator — Phd candidate, Aristotle University of Thessaloniki; Charalambos Karvounis, MD,Phd, Principal Investigator — Professor of Cardiology, School of Medicine, Aristotle University of Thessaloniki; George Giannakoulas, MD,Phd, Principal Investigator — Assistant Professor of Cardiology, School of Medicine, Aristotle University of Thessaloniki; Christos Arvanitidis, Phd, Principal Investigator — Director of Research, Hellenic Center for Marine Research; Ioannis Vizirianakis, PharmD, PhD, Principal Investigator — Associate Professor, School of Pharmacy, Aristotle University of Thessaloniki; James S Michaelson, MD,Phd, Principal Investigator — Associate Professor, Department of Pathology, Harvard Medical School; Kleoniki Keklikoglou, MSc, Principal Investigator — HELLENIC CENTER FOR MARINE RESEARCH; Ivelin Samra, MD, Principal Investigator — Head of cardiology department at MHAT"Hadzy Dimityr" Sliven; Nikolaos Konstantinidis, MD,MSc, Principal Investigator — Phd candidate, Aristotle University of Thessaloniki; Georgios Sofidis, MD,Phd, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- University General Hospital of Thessaloniki AHEPA, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share or not individual participant data with other researchers will depend on the purpose and the scope of the proposed research

REFERENCES:
- [Background] Sianos G, Papafaklis MI, Daemen J, Vaina S, van Mieghem CA, van Domburg RT, Michalis LK, Serruys PW. Angiographic stent thrombosis after routine use of drug-eluting stents in ST-segment elevation myocardial infarction: the importance of thrombus burden. J Am Coll Cardiol. 2007 Aug 14;50(7):573-83. doi: 10.1016/j.jacc.2007.04.059. Epub 2007 Jul 30. PMID 17692740
- [Background] Sianos G, Papafaklis MI, Serruys PW. Angiographic thrombus burden classification in patients with ST-segment elevation myocardial infarction treated with percutaneous coronary intervention. J Invasive Cardiol. 2010 Oct;22(10 Suppl B):6B-14B. PMID 20947930
- [Background] Gibson CM, de Lemos JA, Murphy SA, Marble SJ, McCabe CH, Cannon CP, Antman EM, Braunwald E; TIMI Study Group. Combination therapy with abciximab reduces angiographically evident thrombus in acute myocardial infarction: a TIMI 14 substudy. Circulation. 2001 May 29;103(21):2550-4. doi: 10.1161/01.cir.103.21.2550. PMID 11382722
- [Background] Elgendy IY, Huo T, Bhatt DL, Bavry AA. Is Aspiration Thrombectomy Beneficial in Patients Undergoing Primary Percutaneous Coronary Intervention? Meta-Analysis of Randomized Trials. Circ Cardiovasc Interv. 2015 Jul;8(7):e002258. doi: 10.1161/CIRCINTERVENTIONS.114.002258. PMID 26175531
- [Derived] Karagiannidis E, Papazoglou AS, Sofidis G, Chatzinikolaou E, Keklikoglou K, Panteris E, Kartas A, Stalikas N, Zegkos T, Girtovitis F, Moysidis DV, Stefanopoulos L, Koupidis K, Hadjimiltiades S, Giannakoulas G, Arvanitidis C, Michaelson JS, Karvounis H, Sianos G. Micro-CT-Based Quantification of Extracted Thrombus Burden Characteristics and Association With Angiographic Outcomes in Patients With ST-Elevation Myocardial Infarction: The QUEST-STEMI Study. Front Cardiovasc Med. 2021 Apr 21;8:646064. doi: 10.3389/fcvm.2021.646064. eCollection 2021. PMID 33969012
- [Derived] Karagiannidis E, Konstantinidis NV, Sofidis G, Chatzinikolaou E, Sianos G. Rationale and design of a prospective, observational study for the QUantitative EStimation of Thrombus burden in patients with ST-Elevation Myocardial Infarction using micro-computed tomography: the QUEST-STEMI trial. BMC Cardiovasc Disord. 2020 Mar 11;20(1):125. doi: 10.1186/s12872-020-01393-5. PMID 32160856